CLINICAL TRIAL: NCT03326869
Title: A Prospective Study to Evaluate the Raindrop Near Vision Inlay in Presbyopes Implanted in Corneal Pockets With a Delayed or Non-Delayed Approach
Brief Title: A Study Raindrop Near Vision Inlay in Presbyopes Implanted in Corneal Pockets
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Corneal Inlay supplier no longer in business
Sponsor: Eye Center of North Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECNF17-001
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, multicenter, open label clinical trial where a maximum of 30 non-dominant eyes are implanted with the Raindrop Near Vision Inlay. Each surgical site will be responsible for assigning patients to either the delayed or the non-delayed groupings.
Masking Description: No Masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Delayed (Experimental): Intervention: Raindrop Near Vision Inlay
  In the delayed approach, the corneal pocket is created and dissected but the corneal inlay is not implanted. After one to three months, the corneal inlay is implanted on a second surgical day.
  Interventions: Device: Raindrop Near Vision Inlay
- Non-Delayed (Active Comparator): Intervention: Raindrop Near Vision Inlay
  In the non-delayed approach, the corneal pocket is created and inlay implanted on the same surgical day.
  Interventions: Device: Raindrop Near Vision Inlay

INTERVENTIONS:
Device: Raindrop Near Vision Inlay — The Raindrop Near Vision Inlay was approved by the US FDA in June of 2016 for the improvement of near vision in presbyopic emmetropes. Raindrop is a clear device made of a hydrogel material and resembles a microscopic contact lens; it is the first implantable device that changes the shape of the cornea to correct the refractive errors that cause near vision problems.

SUMMARY:
The objective of this study is to evaluate the Raindrop® Near Vision Inlay for the improvement of near vision in presbyopes implanted in corneal pockets with a delayed or a non-delayed approach.

DETAILED DESCRIPTION:
Patients must be presbyopic with a reading add from +1.5 to +2.5 D, and both emmetropes (MRSE from -0.5 to +0.5 D) as well as ametropes (requiring concurrent LASIK) are included in the investigation. In the non-delayed approach, the corneal pocket is created and inlay implanted on the same surgical day. In the delayed approach, the corneal pocket is created and dissected but the corneal inlay is not implanted. After one to three months, the corneal inlay is implanted on a second surgical day.

ELIGIBILITY:
1.1 Inclusion Criteria:

1.1.1 Patients require a near reading add from +1.5 to +2.5 D in the non-dominant eye.

1.1.2 Patients have a photopic pupil size of at least 3.0 mm in the non-dominant eye.

1.1.3 Patients have a central corneal thickness ≥ 500 microns in the non-dominant eye.

1.1.4 Patients have corrected distance and near visual acuity of 20/25 or better in each eye.

1.1.5 Patients have uncorrected near acuity of 20/40 or worse in the non-dominant eye.

1.1.6 Patients are willing and able to understand and sign a written Informed Consent Form prior to any study-specific procedures.

1.1.7 Patients are willing and able to return for scheduled follow-up examinations for 24 months after corneal inlay implantation.

1.1 Exclusion Criteria:

1.1.1 Patients with clinically significant dry eye (i.e., significant diffuse punctate staining with fluorescein and a tear breakup time less than 8 s) in either eye.

1.1.2 Patients with a planned corneal residual bed thickness that is less than 300 microns (corneal thickness - (intended ablation depth + intended flap thickness)).

1.1.3 Patients with macular pathology based on dilated fundus exam and/or optical coherence tomography (OCT) image.

1.1.4 Patients who would be co-managed by an ophthalmologist or optometrist who is not approved as a ReVision Optics investigator.

1.1.5 Patients with ocular pathology or disease (including pupil pathology such as fixated pupils) that might confound the outcome or increase the risk of adverse event.

1.1.6 Patients taking systemic or topical medications that might confound the outcome or increase the risk of adverse event. Patients taking isotretinoin or amiodarone hydrochloride and any other medication that affects the tear film or accommodation, including but not limited to, mydriatic, cycloplegic and mitotic agents, tricyclic, phenothiazines, benzodiazepines, and first generation antihistamines.

1.1.7 Patients with known sensitivity to any planned study medications. 1.1.8 Patients with residual, recurrent, active or uncontrolled eyelid disease. 1.1.9 Patients with significant corneal asymmetry or irregular topography. 1.1.10 Patients with clinically significant anterior segment pathology. 1.1.11 Patients with any corneal abnormality, including but not limited to, slit lamp findings for corneal staining Grade 3 or higher, recurrent corneal erosion or severe basement membrane disease, and pterygium extending onto the cornea.

1.1.12 Patients with ophthalmoscopic/topographic signs of keratoconus or those who are keratoconus suspect.

1.1.13 Patients with history of Herpes zoster or Herpes simplex keratitis. 1.1.14 Patients with any progressive retinal disease or patients with a history or evidence of retinal vascular occlusion and/or hypercoagulability, because of the risks associated with high pressures during suction application.

1.1.15 Patients with known history of steroid-responsive intraocular pressure increases, glaucoma, preoperative IOP > 21 mm Hg, or are otherwise suspected of having glaucoma.

1.1.16 Patients with amblyopia or strabismus or those who are at risk for developing strabismus postoperatively as determined by corneal light reflex and cover-uncover testing.

1.1.17 Patients with diabetic retinopathy, collagen, vascular, diagnosed autoimmune disease (e.g., lupus, rheumatoid arthritis, fibromylagia), immunodeficiency (e.g., HIV), connective tissue disease, or clinically significant atopic syndrome such as allergies or asthma.

1.1.18 Patients on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing.

1.1.19 Patients with any type of active cancer (ophthalmic or non-ophthalmic). 1.1.20 Patients with uncontrolled infections of any kind. 1.1.21 Patients who are pregnant, lactating, of child-bearing potential and not practicing a medically approved method of birth control, or planning to become pregnant during the course of the trial, and patients with other conditions associated with fluctuation of hormones that could lead to refractive changes.

1.1.22 Patients who actively participate in contact sports (i.e., boxing, martial arts) where impacts to the face and eye are a normal occurrence.

1.1.23 Patients participating in any other ophthalmic or non-ophthalmic drug/device clinical trials during the time of this clinical investigation.

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret L. Fisher, MD, Principal Investigator — Eye Center of North Florida
Locations (1):
- Eye Center of North Florida, Panama City, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed: Intervention: Raindrop Near Vision Inlay
  In the delayed approach, the corneal pocket is created and dissected but the corneal inlay is not implanted. After one to three months, the corneal inlay is implanted on a second surgical day.
  Raindrop Near Vision Inlay: The Raindrop Near Vision Inlay was approved by the US FDA in June of 2016 for the improvement of near vision in presbyopic emmetropes. Raindrop is a clear device made of a hydrogel material and resembles a microscopic contact lens; it is the first implantable device that changes the shape of the cornea to correct the refractive errors that cause near vision problems.
- Non-Delayed: Intervention: Raindrop Near Vision Inlay
  In the non-delayed approach, the corneal pocket is created and inlay implanted on the same surgical day.
  Raindrop Near Vision Inlay: The Raindrop Near Vision Inlay was approved by the US FDA in June of 2016 for the improvement of near vision in presbyopic emmetropes. Raindrop is a clear device made of a hydrogel material and resembles a microscopic contact lens; it is the first implantable device that changes the shape of the cornea to correct the refractive errors that cause near vision problems.
Period: Overall Study
Arm/Group | Delayed | Non-Delayed
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study data has been lost to natural disa | 1 | 1

BASELINE CHARACTERISTICS:
Population: Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed | Non-Delayed | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Visual Acuity
Description: After the inlay procedure, patients will attain functional near acuity in the inlay eye and functional distance vision binocularly.
Time Frame: 24 Months
Population: as for baseline characteristics
Arm/Group | Delayed | Non-Delayed
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Corneal Reaction
Description: Patients implanted with a delayed approach will have minimal incidence of corneal reaction as compared with non-delayed implantation.
Time Frame: 24 Months
Population: as for baseline characteristics
Arm/Group | Delayed | Non-Delayed
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report
Description: Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report
Arm/Group | Delayed | Non-Delayed
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study data has been lost to natural disaster (Hurricane Micheal), therefore there is no study data that is available to report

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT03326869/Prot_001.pdf